CLINICAL TRIAL: NCT06333769
Title: A Phase II Multicenter Clinical Trial of Modified Short-course Radiotherapy Combined With CAPOX and PD-1 Monoclonal Antibody for Locally Advanced Mid-low Rectal Cancer
Brief Title: Modified SCRT Followed by Tislelizumab Plus CAPOX for Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CATIMOR
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Mid-low Rectal Cancer
Keywords: short-course radiotherapy; CAPOX; PD-1 monoclonal antibody
MeSH Terms: interventions — tislelizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Short-course Radiotherapy Combined with CAPOX and Tislelizumab (Experimental): Modified SCRT (GTV 30Gy/5f, CTV 22.5Gy/5f), followed by Tislelizumab and CAPOX q3w *2 cycles. Efficacy and surgery were assessed 2-4 weeks after the end of treatment.
  Interventions: Radiation: Short-course Radiotherapy; Drug: Tislelizumab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Radiation: Short-course Radiotherapy — Rectal lesion + metastatic lymph nodes, GTV 30Gy/5Fx. Pelvic lymphatic drainage area, CTV 22.5Gy/5Fx.
Drug: Tislelizumab — Tislelizumab：200mg，d1，q3w，2 cycles.
Drug: Capecitabine — Capecitabine：1000mg/m2，d1-14，bid, q3w, 2 cycles.
Drug: Oxaliplatin — Oxaliplatin：130mg/m2, d1, q3w, 2 cycles

SUMMARY:
To explore the complete response (CR) rate of modified short-course radiotherapy combined with CAPOX and tislelizumab for locally Advanced Mid-low Rectal Cancer

DETAILED DESCRIPTION:
In the neoadjuvant treatment of rectal cancer, the new mode of short-course radiotherapy and chemotherapy combined with immunotherapy has shown good potential for application. Combining PD-1 antibody with short-course radiotherapy and chemotherapy to increase the tumour-killing and immune-mediated effects of the radiation dose may further improve tumour regression and increase the complete remission rate, providing a promising treatment option for patients with low-grade rectal cancer who are seeking a 'wait-and-see' strategy to preserve organ function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, any gender.
* Pathologically confirmed rectal adenocarcinoma.
* Baseline MR stage T3-4/N+.
* Distance from anal verge ≤12cm.
* No distant metastasis.
* Karnofsky Performance Status ≥70.
* Adequate organ function, no contraindications to surgery, radiotherapy, or immunotherapy.
* Microsatellite/mismatch repair status MSS/pMMR.
* No prior chemotherapy or any other anti-tumor treatment before inclusion.
* No prior immunotherapy.
* Ability to comply with the study protocol during the study period.
* Signed written informed consent.

Exclusion Criteria:

* Pregnant or lactating women.
* Pathological diagnosis of signet ring cell carcinoma.
* History of other malignancies within the past 5 years, except cured skin cancer and cervical carcinoma in situ.
* Uncontrolled epilepsy, central nervous system disorders, or history of psychiatric disorders that, in the opinion of the investigator, may interfere with signing the informed consent form or affect patient compliance with oral medication.
* Clinically significant (i.e., active) cardiac disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) Class II or greater congestive heart failure, or significant arrhythmias requiring drug intervention (see Appendix 12), or history of myocardial infarction within the past 12 months.
* Organ transplant recipients requiring immunosuppressive therapy and long-term steroid users.
* Patients with autoimmune diseases.
* Severe uncontrolled recurrent infections or other severe uncontrolled comorbidities.
* Subjects with baseline hematological and biochemical parameters not meeting the following criteria: hemoglobin ≥90g/L; absolute neutrophil count (ANC) .≥1.5×10^9/L; platelets ≥100×10^9/L; ALT, AST ≤2.5 times the upper limit of normal; ALP ≤2.5 times the upper limit of normal; serum total bilirubin <1.5 times the upper limit of normal; serum creatinine <1 times the upper limit of normal; serum albumin ≥30g/L.
* Known deficiency of dihydropyrimidine dehydrogenase (DPD).
* Allergy to any investigational drug components.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) rate | From enrollment to 3 month and during follow-up
  Including pCR and CCR.

SECONDARY OUTCOMES:
Organ preservation rate | 1 year.
  Sphincter-saving rate in enrolled patients
Quality of life | Before each treatment, before surgery and during follow-up.
  EORTC Core Quality of Life questionnaire (QLQ-C30)，range from 0-100, with comprehensive assessment indicators, including positive and negative indicators.
3y-DFS | From enrollment to 36 month
3-year OS | From enrollment to 36 month
  The percentage of patients enrolled who are still alive three years after their initial enrollment.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The Second Hospital of Longyan, Longyan, Fujian
  - Jinjiang Municipal Hospital, Quanzhou, Fujian